CLINICAL TRIAL: NCT06264973
Title: Maternal and Fetal/Neonatal Pharmacokinetics and - Dynamics of Corticosteroids During Pregnancy as Treatment for Fetal Lung Maturation MaDyCo-study
Brief Title: Maternal and Fetal/Neonatal Pharmacokinetics and - Dynamics of Corticosteroids During Pregnancy
Acronym: MaDyCo
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Sam Schoenmakers, Gynaecologist, perinatologist, Erasmus Medical Center
Other Study IDs: NL9318
Record Dates: First submitted 2023-07-04; First posted 2024-02-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Improving pregnancy outcome is essential in improving health of both parents and their offspring during the life course. Preterm birth (PTB) occurs in 10-15% of all pregnancies, is the leading cause of perinatal mortality and morbidity {Goldenberg, 2008}, has long-term adverse consequences for postnatal health {Huddy, 2001} and is a burden for health care expenditure. In order to improve neonatal outcome, antenatal corticosteroids (ACS) are routinely administered to women at risk for preterm delivery before 34 weeks of pregnancy. {Jobe, 2018;Roberts, 2017;Travers, 2018} However, the current, worldwide standard of care, for the use of ACS is still based on animal experiments performed in the 1970's. {Liggins, 1969} Although ACS treatment to improve neonatal outcome was clinically introduced in the 70's, still only two dosing regimens are used, neither of which have been investigated, re-evaluated or refined to determine the optimal doses or treatment interval. With the current health care approach of personalized medicine in mind, the same universal approach for everybody, independent of gestational age, number of fetus, maternal weight or comorbidity one dose does not fit all since it often has not the desired effect. Due to the lack of optimization of the above mentioned synthetic corticosteroid drug regimens {Kemp, 2019}, significant gaps in knowledge exist. An important aspect to set up, investigate and understand dosing and also dosing interval experiments, is knowledge of the maternal individual pharmacokinetics and pharmacogenetics of the drug of interest during pregnancy.

DETAILED DESCRIPTION:
A clinical observational study will be performed in women admitted at the Department of Obstetrics at the Sophia Children's Hospital/Erasmus MC for suspicion of preterm birth with a gestational age of 23+5 weeks until 33+6 weeks. Antenatal corticosteroids will be administered according to the local standard protocol (12 mg betamethasone intramuscular with a 24 hours intervall). Importantly, clinical management of women with suspicion of preterm birth will not be affected by the proposed study. After inclusion, repetitive blood sampling according to the following schedule: t0 (administration), t0-30 min, t10-12hrs and t20-24 hrs. Umbilical cord will be sampled directly after birth as fetal determinant in which corticosteroids and their metabolites will be measured. Also, neonatal blood samples (drawn by the paediatricians as part of standard care) will be used for measurement of corticosteroids and their metabolites. Maternal blood samples will furthermore be analysed for determinants effecting pharmacokinetics such as oestradiol.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years of age.
2. Admitted at the Department of Obstetrics at Erasmus MC - Sophia for suspicion of preterm birth with a gestational age of 23+5 weeks until 33+6 weeks.
3. Understanding of Dutch in speaking and reading.
4. Written informed consent.

   In order for the neonate to be able to participate in this study, the parent must meet the following criteria:
5. Older than 18 years of age.
6. Admitted at the Department of Obstetrics at Erasmus MC - Sophia for suspicion of preterm birth with a gestational age of 23+5 weeks until 33+6 weeks.
7. Understanding of Dutch in speaking and reading.
8. Written informed consent for the neonate.

Exclusion Criteria:

1. Women unable or unwilling to agree with the procedures.
2. Women unable or unwilling to give written informed consent.
3. Women with acute obstetric complications requiring immediate delivery at time of admission.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: Pregnant women admitted at the Department of Obstetrics at Erasmus MC - Sophia for suspicion of preterm birth with a gestational age of 23+5 weeks until 33+6 weeks. Postpartum, the neonates will also be included in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics of antenatal corticosteroids by investigation of betamethasone concentrations in serum using mmol/l | 2 days
  To examine the pharmacokinetics in maternal blood of standard regimen at the Erasmus MC of two doses of 12 mg betamethasone intramuscular with a 24 hours interval

SECONDARY OUTCOMES:
Maternal age | 2 days
  To examine the relation between maternal age and the pharmacokinetics of the primary objective
Fetal sex | 2 days
  To examine the relation between fetal sex and the pharmacokinetics of the primary objective
Maternal weight/BMI in kg and kg/m2 | 2 days
  To examine the relation between maternal weight/BMI and the pharmacokinetics of the primary objective
Number of fetus | 2 days
  To examine the relation between the number of fetus and the pharmacokinetics of the primary objective
Parity: the number of times a woman has given birth to a live neonate (any gestation) or at 24 weeks or more | 2 days
  To examine the relation between parity the pharmacokinetics of the primary objective
PE by urine measurement of protein-creatinine ratio | 2 days
  To examine the relation between pre-eclampsia and the pharmacokinetics of the primary objective
Oestradiol concentration in serum in mmol/l | 2 days
  To examine the relation between oestradiol on pharmacokinetics of the primary objective
Cord blood and neonatal blood concentration in mmol/l of corticosteroids | Delivery
  To examine the relation between pharmacokinetics in cord blood and neonatal blood

OTHER OUTCOMES:
CYP3A4 level | 2 days
  To examine the relation between CYP3A4 genotype and the pharmacokinetics of the primary objective

CONTACTS AND LOCATIONS:
Overall Officials: Sam Schoenmakers, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided